CLINICAL TRIAL: NCT00700895
Title: A Randomized Controlled Trial to Assess the Clinical Benefits of a Pharmacogenetics-Guided Dosing Regimen for Calculating Warfarin Maintenance Dose
Brief Title: Assessing the Clinical Benefits of a Pharmacogenetics-Guided Dosing Regiment for Calculating Warfarin Maintenance Dose
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Haematology-Oncology, Dr. Goh Boon Cher, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PG01/11/06
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Indications for Warfarin Therapy
MeSH Terms: interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pharmacogenetics-guided dosing group (Experimental): For patients randomized to the pharmacogenetics-guided dosing group, this 10mls of blood will be immediately sent for genotyping studies. Genotyping results will be available for pharmacogenetics-guided dosing within 3 working days, (ranging 3 to 5 days). During this period, if patients need to be initiated on anticoagulation, a low molecular weight heparin, Fraxiparine, will be given. Fraxiparine will be overlapped with warfarin for 2 to 3 days until target INR is achieved. Elective cases should have the pharmacogenetics-based warfarin dose available at the time of warfarin therapy.
  Interventions: Drug: Warfarin Sodium
- Traditional dosing group (Experimental): For patients randomized to the traditional dosing regime, the blood will be stored and genotyped retrospectively at the end of the study. Overlapping of warfarin with Fraxiparine or heparin till target INR is achieved is allowed for this group as per normal clinical practice. All warfarin dosage adjustments based on INR results will be according to the current protocol used by the NUH Anticoagulant Clinic.
  Interventions: Drug: Warfarin Sodium

INTERVENTIONS:
Drug: Warfarin Sodium — All predicted warfarin dose will be administered by rounding down to the nearest 0.5 mg. Warfarin (Marevan®) is available as 1mg (brown), 3 mg (blue) and 5 mg (pink) oral tablets from GlaxoSmithKline Pte. Ltd.
  Other Names: Warfarin (Marevan®)

SUMMARY:
Interethnic differences in warfarin dose requirements in the Asian population have been well described. Our previous studies showed that warfarin maintenance doses in our multi-ethnic population were closely related to patient demographics and genetic polymorphisms in cytochrome(CYP)P4502C9 and vitamin K epoxide reductase complex subunit 1(VKORC1). A retrospective regression model combining these predictors accounts for 57.8% of the variability in warfarin dose.

DETAILED DESCRIPTION:
Hypothesis: We hypothesize that warfarin dose requirement could be more accurately predicted using a simplified genotyping procedure requiring the identification of a single CYP2C9 allele and a single nucleotide polymorphism of VKORC1 to discern between the 2 major haplotypes H1 and H7.

Aims: The aim is to compare the clinical benefits of genetics-guided dosing versus traditional trial and error dosing with protocol guided-adjustments. Two secondary objectives are (1) to prospectively evaluate a dosing algorithm built on demographics and genetic predictors; (2) to assess the feasibility of a simplified test for CYP2C9*3 and VKORC1 SNP in clinical practice.

Methodology: A randomized controlled trial targeted at accruing 100 patients with indication for wafarin therapy. The endpoint for comparing genetics-guided dosing against traditional dosing method at the anticoagulant clinic is the number of dosage titrations to achieve targeted International Normalized Ratio (INR) at 1, 2 and 3 months of initializing warfarin. Upon reaching steady-state, pharmacokinetics of warfarin R- and S-isomers will be assessed for correlation with dose requirements based. An assay for easy identification of genetic polymorphisms required in this dosing regimen in a clinic setting will also be validated.

Significance: This concerted, multi-disciplinary effort to bring pharmacogenetics-based therapy from bench to bedside has the potential to reduce the efforts incurred with multiple dose titrations of the most commonly prescribed oral anticoagulant. With the aid of mathematical modeling, a simplified and more cost-effective genotyping method could be implementation for the future treatment and prophylaxis of thromboembolic diseases.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. New indication for warfarin therapy
3. No previous history of liver disease; transaminases must be less than 3 times upper limit of normal and bilirubin within normal range
4. No previous history of malabsorption syndrome or chronic diarrheal conditions
5. Written, informed consent

Exclusion Criteria:

1. Uncontrolled hypertension
2. Peptic ulcer disease
3. Any other medical conditions as deemed unfit for warfarin therapy based on clinical judgement of primary physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2006-08; Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
No. of dosage titrations required to achieve targeted INR at 3 months of initializing warfarin. | 3 months
  1. Number of dosage titrations/adjustments required to achieve targeted International Normalized Ratio (INR) at 3 months of initializing warfarin. The number of titrations refers to the number of times warfarin dosage was adjusted when INR was out of target range (>1.9 and ≤ 3.1) or in response to an adverse event or therapeutic failure. This endpoint will be compiled every 4 weeks, up to 3 months after the initialization of warfarin therapy

SECONDARY OUTCOMES:
pharmacokinetics of warfarin R- and S-enantiomers | 3 months
  Upon reaching steady-state, pharmacokinetics of warfarin R- and S-enantiomers will be determined for correlation with dose requirements and genotypes based on a single 5ml blood sample taken after achieving target INR without a change in dose for at least 3 months. Warfarin concentrations will be measured using a validated method through a high-performance liquid chromatography (HPLC) method modified from Henne et al.

CONTACTS AND LOCATIONS:
Overall Officials: Boon Cher Goh, MBBS, MRCP, Principal Investigator — National University Hospital, Singapore
Locations (2):
- University of Malaya Medical Centre, Kuala Lumpur, Malaysia
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Wong HJ, Teo YN, Teo YH, Syn NL, Wong AL, Teoh HL, Seet RCS, Lee SC, Goh BC, Sia CH. Subgroup analysis of genotype guided vs traditional warfarin dosing in Asian patients from an open label randomized trial. Sci Rep. 2026 Jan 2;16(1):3670. doi: 10.1038/s41598-025-33831-9. PMID 41484425
- [Derived] Syn NL, Wong AL, Lee SC, Teoh HL, Yip JWL, Seet RC, Yeo WT, Kristanto W, Bee PC, Poon LM, Marban P, Wu TS, Winther MD, Brunham LR, Soong R, Tai BC, Goh BC. Genotype-guided versus traditional clinical dosing of warfarin in patients of Asian ancestry: a randomized controlled trial. BMC Med. 2018 Jul 10;16(1):104. doi: 10.1186/s12916-018-1093-8. PMID 29986700